CLINICAL TRIAL: NCT06768203
Title: The Effect of Umbilical Vein Catheterization on Splanchnic Oxygenation
Brief Title: The Effect of Umbilical Vein Catheterization on Splanchnic Oxygenation in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ozge Surmeli Onay, Professor Doctor, Eskisehir Osmangazi University
Other Study IDs: EskisehirOU-UVC STUDY
Record Dates: First submitted 2024-12-23; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Feeding Intolerance; Necrotising Enterocolitis Neonatal
Keywords: umbilical venous catheter; splanchnic oxygenation; near-infrared spectroscopy; small for gestational age; feeding intolerance
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The UVC (+) Study Group: Infants who indicated UVC placement, and for whom NIRS measurements were taken both before and after UVC placement were included in the UVC (+) Study Group.
  Interventions: Other: umbilical vein catheterization
- The UVC (-) Control Group: Infants who did not have a UVC but matched the Study Group regarding gestational age and birth weight constituted the UVC (-) Control Group.
  Interventions: Other: Control

INTERVENTIONS:
Other: umbilical vein catheterization — In our NICU, UVC placement is a sterile bedside procedure carried out by pediatric residents, neonatology fellows, and neonatology specialists, using polyurethane, single-lumen catheters sized according to the infant's weight: 3.5 Fr for those under 1500 g and 5 Fr for those over 1500 g. Catheter placement is performed using the Modified Shukla-Ferrara Formula
  Groups: The UVC (+) Study Group
Other: Control — No umbilical vein catheter was inserted in these infants.
  Groups: The UVC (-) Control Group

SUMMARY:
Objectives: This study aimed to assess the impact of umbilical vein catheter (UVC) placement on splanchnic oxygenation in preterm infants.

Methods: In our single-center, prospective, observational cohort study, near-infrared spectroscopy probes were placed to monitor regional splanchnic oxygen saturation (rSO2S) and calculate fractional tissue oxygen extraction (FOE) in preterm infants (GA < 34 weeks, BW 1000-2000 g) for one week post-stabilization. Gestational age-matched UVC (+) and (-) Groups were clinically and physiologically compared, before and after UVC placement/removal.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate how the insertion of an umbilical vein catheter (UVC) affected the splanchnic oxygenation of preterm newborns..

ELIGIBILITY:
Inclusion Criteria:

* Parents agreed to participate in the study
* Infants born in our hospital, who were followed up in the NICU, with a gestational age of <34 weeks and a birth weight of 1000-2000 grams
* Infants who indicated UVC placement, and for whom NIRS measurements were taken both before and after UVC placement were included in the UVC (+) Study Group
* Infants who did not have a UVC but matched the Study Group regarding gestational age and birth weight constituted the UVC (-) Control Group

Exclusion Criteria:

* Infants who died during the first week of life
* Transferred to another hospital
* Chromosomal anomalies
* Major congenital anomalies affecting splanchnic bed monitoring (such as congenital heart disease, abdominal wall defects, or congenital diaphragmatic hernia)
* Inherited metabolic disorders
* Hydrops fetalis
* TORCH infections
* Multiple organ failure
* Spontaneous intestinal perforation
* Lesions in the area where the NIRS sensor was placed
* If UVC was removed for any reason before 24 hours
* Severe anemia or polycythemia (Infants with a birth hemoglobin (Hb) level of 10 g/dl or below were considered severe anemic, and those with a Hb level of 22 g/dl or above were considered polycythemic)

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants whose gestational age is <34 weeks, birth weight 1000-2000 grams.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
The splanchnic oxygenation (rSO2S) | first week of life (7 days)
  The primary outcomes included comparing continuously recorded rSO2S and FOE values during the first week of life between the UVC (+) and UVC (-) groups, assessing rSO2S and FOE measurements within the UVC (+) Group before and after UVC placement and removal, and determining the impact of UVC on splanchnic oxygenation

SECONDARY OUTCOMES:
The incidence of feeding intolerance and necrotizing enterocolitis. | During hospital stay (maximum 3 months)
  The secondary outcomes involve evaluating the relationship between UVC presence and the incidence of feeding intolerance and necrotizing enterocolitis.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Surmeli Onay, Study Director — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van der Heide M, Dotinga BM, Stewart RE, Kalteren WS, Hulscher JBF, Reijneveld SA, Bos AF, Kooi EMW. Regional splanchnic oxygen saturation for preterm infants in the first week after birth: reference values. Pediatr Res. 2021 Oct;90(4):882-887. doi: 10.1038/s41390-020-01323-3. Epub 2021 Jan 27. PMID 33504960
- [Result] Surmeli Onay O, Velipasaoglu M, Tutal M, Sarilar TD, Cakil Saglik A, Bilgin M, Aydemir O, Barsan Kaya T, Tanir HM, Tekin AN. The effect of drip versus intermittent feeding on splanchnic oxygenation in preterm infants with intrauterine growth restriction: a prospective randomized trial. Eur J Pediatr. 2023 Mar;182(3):1317-1328. doi: 10.1007/s00431-023-04810-x. Epub 2023 Jan 13. PMID 36637540
- [Result] Sulemanji M, Vakili K, Zurakowski D, Tworetzky W, Fishman SJ, Kim HB. Umbilical Venous Catheter Malposition Is Associated with Necrotizing Enterocolitis in Premature Infants. Neonatology. 2017;111(4):337-343. doi: 10.1159/000451022. Epub 2017 Jan 17. PMID 28092913

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT06768203/Prot_SAP_000.pdf